CLINICAL TRIAL: NCT06438601
Title: A Clinical Comparison of Two Multifocal Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-159
Record Dates: First submitted 2024-05-24; First posted 2024-06-03 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-05

CONDITIONS: Astigmatism; Presbyopia
MeSH Terms: conditions — Astigmatism; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (omafilcon A) (Experimental): All participants will wear lens A for 15 minutes (Period 1).
  Interventions: Device: Lens A (omafilcon A)
- Lens B (comfilcon A) (Experimental): All participants will wear lens B for 15 minutes (Period 2).
  Interventions: Device: Lens B (comfilcon A)

INTERVENTIONS:
Device: Lens A (omafilcon A) — 15 minutes of daily wear.
  Arms: Lens A (omafilcon A)
Device: Lens B (comfilcon A) — 15 minutes of daily wear.
  Arms: Lens B (comfilcon A)

SUMMARY:
This study aims to compare the short-term clinical performance of the two study contact lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the short-term clinical performance of two multifocal toric soft contact lenses after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged 35 years or over and have capacity to volunteer.
2. They understand their rights as a subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They agree not to participate in other clinical research for the duration of this study.
5. They are currently wearing soft contact lenses or have done so within the past 12 months.
6. They have a spherical prescription between +10.00 and -10.00DS inclusive, (based on the ocular refraction).
7. They have astigmatism of between -0.75 and -5.75DC (based on the ocular refraction) in each eye.
8. They have a reading addition component to their spectacle refraction of between +0.75 and +2.50DS.
9. They can be satisfactorily fitted with the study lenses.
10. They own a wearable pair of spectacles.

Exclusion Criteria:

1. They have an ocular disorder which would normally contraindicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medications such as eye drops or ointment.
4. They have had cataract surgery.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
8. They have eye or health conditions including immunosuppressive or infectious diseases which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.
9. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codina, PhD,MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty participants were screened. Of those, four participants were ineligible and excluded from the study. Thirty-six participants were enrolled.
Groups:
- Lens A (Omafilcon A): All participants wore Lens A for 15 minutes (Period 1).
  Lens A (omafilcon A): 15 minutes of daily wear.
- Lens B (Comfilcon A): All participants wore Lens B for 15 minutes (Period 2).
  Lens B (comfilcon A): 15 minutes of daily wear.
Period: Period 1: Lens A (15 Minutes)
Arm/Group | Lens A (Omafilcon A) | Lens B (Comfilcon A)
Started | 36 | 0 (All participants received Lens A in Period 1.)
Completed | 34 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Use of eye drops between study visits | 1 | 0
Period: Period 2: Lens B (15 Minutes)
Arm/Group | Lens A (Omafilcon A) | Lens B (Comfilcon A)
Started | 0 (All participants received Lens B in Period 2.) | 34
Completed | 0 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all enrolled participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Four participants were ineligible, of which two were ineligible due to astigmatism in their left eye, one had poor visual acuity in their right eye and one did not require a reading add.
  Participants
    Female | 23
    Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Distance Vision
Description: Subjective Distance Vision will be measured on a scale from 0-100 (Where 0= Extremely poor. Intolerable. Lenses cannot be worn. 100= Excellent. Unaware of any visual loss).
Time Frame: At the end of 15 minutes of daily wear
Population: All participants that completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lens A (Omafilcon A) | Lens B (Comfilcon A)
Number analyzed (Participants) | 34 | 34
units on a scale | 77.1 (19.6) | 80.0 (14.5)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately sixteen weeks.
Description: The Adverse Events cannot be attributed to one intervention or the other. Therefore, an additional Arm/Group was added to report these Adverse Events (i.e., a total of 3 Arms/Groups).
Groups:
- Lens A (Omafilcon A): Participants that received Lens A
- Lens B (Comfilcon A): Participants that received Lens B
- No Intervention: All Study Participants
Arm/Group | Lens A (Omafilcon A) | Lens B (Comfilcon A) | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 2/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens A (Omafilcon A) (N=36) | Lens B (Comfilcon A) (N=34) | No Intervention (N=36)
Suspect vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study lenses.
Sub-conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study lenses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT06438601/Prot_SAP_000.pdf